CLINICAL TRIAL: NCT04971915
Title: The Effect of Minimalist Footwear on the Anthropometric and Biomechanical Parameters of the Lower Limb and Foot During Long-Term Wearing: A Randomized Clinical Trial
Brief Title: The Effect of Minimalist Footwear on the Anthropometric and Biomechanical Parameters of the Lower Limb and Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Zdenek Svoboda, Assistent Professor, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IGA_FTK_2021_010
Record Dates: First submitted 2021-07-05; First posted 2021-07-22 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Footwear
Keywords: minimalist footwear; shoes; biomechanics; anthropometric parameters; foot; walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimalist footwear (Experimental): The participants in the experimental group will receive one pair of minimalist footwear and will be asked to use them for the interventional period.
  Interventions: Other: minimalist footwear
- control (No Intervention): The participants in the control group will be asked to wear their standard footwear as before participating in the study.

INTERVENTIONS:
Other: minimalist footwear — The intervention consists of wearing the minimalist footwear in recommended progression during the interventional period (6months). The intial load starts at 2,500 steps a day and will be gradually increased up according to the participant´s tolerance rate to the footwear wearing to fully use over the final period. Participants are instructed to report all issues and difficulties possibly connected to the intervention. There will be the opportunity to consult any issue connected with footwear or their wearing through the duration of the research.
  Arms: minimalist footwear

SUMMARY:
The study aims to determine whether 6months of wearing minimalist footwear causes changes in anthropometric parameters of the foot and the biomechanical parameters of the foot and lower limb.

DETAILED DESCRIPTION:
The minimalist footwear represents an alternative style of footwear wearing, which could allow the foot to move more naturally compared to the footwear wearing in conventional footwear. That footwear is characterized by no cushioning, wide toe box, zero foot drop, thin sole (1,5 - 8 mm), low weight, and high flexibility of footwear. This study aims to determine the effect of 6months of wearing minimalist footwear on the foot and lower limb's anthropometric and biomechanical parameters.

The study is designed as a parallel interventional study. The sample size consists of 50 healthy individuals divided into experimental and control groups by randomization. All participants undergo the initial examination and baseline and final measurement focused on the foot anthropometry and kinetics and kinematics of the foot and lower limb during walking. Besides, the experimental group undergoes a 6months intervention of wearing minimalist footwear, during which the participants will record their movement behavior by electronic diary.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Individuals without previous experience in wearing minimalist footwear

Exclusion Criteria:

* Significant deformities of the feet and toes
* Pain of the musculoskeletal system
* Injury, congenital or gained defect of the musculoskeletal or neural system in past
* Undergo operation of lower limbs in past or during research

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Change in range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle | at baseline and at the end of 6 months intervention
  Range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in maximal value of range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle | at baseline and at the end of 6 months intervention
  Maximal value of range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in minimal value of range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle | at baseline and at the end of 6 months intervention
  Minimal value of range of motion of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in angular velocity of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle | at baseline and at the end of 6 months intervention
  Angular velocity of pelvis, joints of lower limb and foot in coronal, transversal and frontal plane during stance phase of the gait cycle will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in walking velocity | at baseline and at the end of 6 months intervention
  Walking velocity will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in walking cadence | at baseline and at the end of 6 months intervention
  Walking cadence will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in step length during walking | at baseline and at the end of 6 months intervention
  Step length will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in duration of stance phase of the gait cycle | at baseline and at the end of 6 months intervention
  Duration of stance phase of the gait cycle will be measured by the Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in maximum value of the vertical component of ground reaction force during walking | at baseline and at the end of 6 months intervention
  Maximum value of the vertical component of ground reaction force will be measured by two force plates Kistler (Kistler, Winterhur, Switzerland) synchronized with Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in minimum value of the vertical component of ground reaction force during walking | at baseline and at the end of 6 months intervention
  Minimum value of the vertical component of ground reaction force will be measured by two force plates Kistler (Kistler, Winterhur, Switzerland) synchronized with Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in impulse of the vertical component of ground reaction force during walking | at baseline and at the end of 6 months intervention
  Impulse of the vertical component of ground reaction force will be measured by two force plates Kistler (Kistler, Winterhur, Switzerland) synchronized with Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in lower limbs joints moments during walking | at baseline and at the end of 6 months intervention
  Lower limbs joints moments will be measured by two force plates Kistler (Kistler, Winterhur, Switzerland) synchronized with Vicon Vantage V5 (Vicon Motion System, London, Great Britain).
Change in peak plantar pressure at anatomical regions of the foot sole during walking | at baseline and at the end of 6 months intervention
  Peak plantar pressure at anatomical regions of the foot sole during walking will be measured by pressure plate 2M footscan® (RSscan International NV, Paal, Belgium).
Change in contact time at anatomical regions of the foot sole during walking | at baseline and at the end of 6 months intervention
  Contact time at anatomical regions of the foot sole during walking will be measured by pressure plate 2M footscan® (RSscan International NV, Paal, Belgium).
Change in contact area at anatomical regions of the foot sole during walking. | at baseline and at the end of 6 months intervention
  Contact area at anatomical regions of the foot sole during walking will be measured by pressure plate 2M footscan® (RSscan International NV, Paal, Belgium).
Change in pressure-time integral at anatomical regions of the foot sole during walking | at baseline and at the end of 6 months intervention
  Pressure-time integral at anatomical regions of the foot sole during walking will be measured by pressure plate 2M footscan® (RSscan International NV, Paal, Belgium).
Change in maximum force at anatomical regions of the foot sole during walking | at baseline and at the end of 6 months intervention
  Maximum force at anatomical regions of the foot sole during walking will be measured by pressure plate 2M footscan® (RSscan International NV, Paal, Belgium).
Change in foot length | at baseline and at the end of 6 months intervention
  Foot length will be measured by RSS 3D Scanner (RSScan International NV, Paal, Belgium).
Change in foot width | at baseline and at the end of 6 months intervention
  Foot width will be measured by RSS 3D Scanner (RSScan International NV, Paal, Belgium).
Change in tactile-foot perception | at baseline and at the end of 6 months intervention
  Tactile-foot perception will be measured by Baseline Tactile Monofilaments (Fabrication Enterprises, White Plains, NY, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Lenka Murinova, Study Director — Faculty of Physical Culture, Palacky University Olomouc
Locations (2):
- Czechia (2):
  - Faculty of Physical Culture, Palacky University Olomouc, Olomouc
  - Palacky University Olomouc, Faculty of Physical Culture, Olomouc

IPD SHARING:
Plan to Share IPD: No